CLINICAL TRIAL: NCT04400448
Title: Acceptance of Telemedicine in Outpatient Clinic Consultations During COVID-19 Pandemic. An International, Cross-sectional Study
Brief Title: Acceptance of Telemedicine During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Luis Sánchez Guillen, Colorectal Surgeon Hospital General Universitario Elche, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: TELECOVID
Record Dates: First submitted 2020-05-14; First posted 2020-05-22 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Covid-19
Keywords: telemedicine; patient acceptance; covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, due to the effects of COVID-19 pandemic, there is an imperative need to change the healthcare model. In this regard, telemedicine has proved very useful in health crises, in which there is a possibility of infection between people, offering remote access to medical care. Telemedicine has been used in many chronic diseases such as asthma and chronic obstructive pulmonary disease, diabetes mellitus, and appears to be well accepted by patients. However, few studies have been conducted in surgical services and in other diseases. Therefore, the aim of this study is to assess the level of acceptance of the patients, in this pandemic situation, to a telemedicine follow-up in different departments.

This is an observational, cross-sectional, multicenter and international study with prospective and retrospective data collection. To evaluate patients' acceptance, we used the validated questionnaire Telehealth usability questionnaire (TUQ). In addition, all patients will provide an overall satisfaction score for telemedicine on a scale from 1 to 5 (1=lowest; 5=highest satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Patients contacted by telemedicine (phone and/or video call) during the COVID-19 pandemic in outpatient clinics
* Follow-up of patients with any chronic disease and postoperative patients, preoperative and urgent consultation
* Age greater than or equal to 18 years

Exclusion Criteria:

* Patients with cognitive or sensory difficulties or with insufficient comprehension of the language in which the survey is conducted
* Patients who decline to take part in the telephone survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who met the described inclusion criteria will be included in the registry. Participants will be asked to answer an anonymous and voluntary questionnaire by telephone, that will be completed online by the researcher and collaborators through a Google form, aimed to assess the acceptance of the use of telemedicine in consultations during the pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Acceptance of telemedicine | 1 month
  Acceptance of telemedicine in consultations during the COVID-19 pandemic. To evaluate patients' acceptance, we used the validated questionnaire Telehealth usability questionnaire (TUQ) as a model. The resulting questionnaire has 10 questions.

SECONDARY OUTCOMES:
Patient satisfaction | 1 month
  Global satisfaction score on a scale from1 to 5 (1=lowest; 5=highest satisfaction)

IPD SHARING:
Plan to Share IPD: Undecided